CLINICAL TRIAL: NCT03277859
Title: Strength and Awareness in Action: an Intervention for Post-Acute TBI Headaches (SAA-TBI)
Acronym: SAA-TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Lisa Brenner, Director of Rocky Mountain Mental Illness, Research, Education and Clinical Center, VA Eastern Colorado Health Care System
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 17-0785
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Traumatic Brain Injury; Post-concussive Headaches
Keywords: Yoga; Veterans; Traumatic Brain Injury; Post-concussive Headaches; Post-concussive Symptoms
MeSH Terms: conditions — Brain Injuries, Traumatic; Post-Concussion Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be block randomized in a stratified manner to SAA-TBI or a waitlist using a 1:1 ratio. The waitlist group will initially receive 8 weeks of enhanced treatment as usual (ETU).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YOGA-NOW (Experimental): Participant will start the SAA-TBI (yoga) about 2 weeks (+/- 2 weeks) after Study Visit 3.
  Interventions: Behavioral: SAA-TBI
- YOGA-WAIT (Active Comparator): Participant will start SAA-TBI (yoga) about 10 weeks (+/- 2 weeks) after Study Visit 3.
  Interventions: Behavioral: SAA-TBI

INTERVENTIONS:
Behavioral: SAA-TBI — Yoga twice a week for 75 minutes for 8 weeks

SUMMARY:
The specific aims of the proposed study are to evaluate: 1) the feasibility of design elements of a Strength and Awareness in Action: an Intervention for Post-Acute TBI Headaches (SAA-TBI) intervention trial (e.g., an exercise run-in to facilitate participant retention); 2) yoga instructor fidelity; and 3) variability estimates for candidate proximal and distal outcomes. Performance of validated measures, including those associated with quality of life, as well as data collected via ecological momentary assessment and pedometry (physical activity) will be evaluated.

DETAILED DESCRIPTION:
A signature injury being sustained by Veterans from recent conflicts is mild traumatic brain injury (mTBI). For some, this condition is associated with multiple disabling post-concussive symptoms, including post-concussive headaches (PCH). PCHs are notoriously resistant to medication alone, and are associated with increased muscle tension, avoidance of physical activities, and anxiety related to having chronic pain. In this study, the feasibility (ease of implementation) of the design elements of an interventional trial of Strength and Awareness in Action: an Intervention for Post-Acute TBI Headaches (SAA-TBI) will be explored. Yoga is operationalized as a practice involving physical postures, breath awareness, breathing exercises and mindfulness meditation. It is conceptualized as having three "active ingredients" (i.e., regulation of the autonomic nervous system via physical activity/breathing exercises, release of muscular tension associated with headaches, and mindfulness/acceptance). The specific aims of the proposed study are to evaluate: 1) the feasibility of design elements of an SAA-TBI intervention trial (e.g., an exercise run-in to facilitate participant retention); 2) yoga instructor fidelity; and 3) variability estimates for candidate proximal and distal outcomes. Performance of validated measures, including those associated with quality of life, as well as data collected via ecological momentary assessment and pedometry (physical activity) will be evaluated. Project aims will be evaluated using an experimental design where participants will be block randomized in a stratified manner to SAA-TBI or a waitlist using a 1:1 ratio. The waitlist group will initially receive 8 weeks of enhanced treatment as usual (ETU). The participants in the waitlist condition will be offered SAA-TBI, after the initial group has completed the intervention. Both groups of participants will complete multiple measures at baseline and after the conclusion of the intervention. Maintenance among the intervention group will also be explored. Participants will be asked to complete daily homework documenting their headaches and yoga practice outside of class, and be provided with multiple modalities (web-based, mobile app, text, or paper and pencil) by which this can be accomplished. In specific, the proposed study will evaluate the feasibility of the trial design for an accessible, non-pharmacological, yoga-based intervention for chronic PCH pain among Veterans with mTBI, with the long-term goal of informing future efficacy trials.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 55
* Able to provide informed consent
* History of mTBI per the Ohio State University TBI-ID (OSU-TBI-ID)
* History of PCH pain (TTH, migraine, or mixed), with onset of pain or increase in previous headache pain having occurred within one month of mTBI as determined by structured examination using criteria outlined in the International Classification of Headache Disorders-3 beta (ICHD-3 beta)
* Duration of PCH pain being greater than one year as determined by structured medical examination
* Score of >49 on the Headache Impact Test-6 (HIT-6)
* Medical clearance by study provider to participate in yoga protocol

Exclusion Criteria:

* Younger than 18, or older than 55 years of age
* Active substance dependence, excluding Cannabis dependence (based on local issues regarding the legality of cannabis), as determined by structured clinical interview
* Moderate to severe TBI as determined per the OSU-TBI-ID
* Identification of active psychosis as determined by structured clinical interview
* Failing to receive medical clearance by study provider;
* Inability to participate in the manualized intervention without postures being significantly modified
* Already participating in an ongoing consistent yoga practice (two or more times weekly)
* Involvement in another research interventional trial aimed at addressing pain-related symptoms.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Headaches per week | Change from baseline to approximately 20 weeks
  Headache Tracking Form (HTF) will query about daily headache frequency, duration, severity, and treatment per event.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Brenner, PhD, Principal Investigator — VA Eastern Colorado Health Care System
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, Colorado, United States